CLINICAL TRIAL: NCT06233331
Title: Phase I Dose Escalation Study of the Use of ACU-D1, a Topical Proteasome Inhibitor in HPV Associated Vulvar and Perianal Lesions in People With HIV
Brief Title: Use of ACU-D1 in HPV Associated Vulvar and Perianal Lesions in People With HIV
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Georgia Center for Oncology Research & Education (Other)
Responsible Party: Principal Investigator, Lisa Flowers, Professor, Emory University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006195
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Human Papilloma Virus; Human Immunodeficiency Virus; Anal Intraepithelial Neoplasia; High-Grade Squamous Intraepithelial Lesions
Keywords: HIV; HPV; Anal Intraepithelial Neoplasia
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Squamous Intraepithelial Lesions

STUDY DESIGN:
Intervention Model Description: This study utilizes a dose escalation phase across a total of 3 dose escalation levels using a standard 3+3 design. Initial three study participants will be enrolled in Dose Level 1 for 4 weeks. If there are no dose-limiting toxicities (DLTs) then 3 new study participants will proceed to Dose level 2. If these 3 study participants do not demonstrate any DLTs then the last 3 study participants will proceed to Dose level 3 for 4 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Level 1 (Experimental): Initial three study participants will be enrolled in Dose Level 1, 2.5% ACU-D1 twice daily for 4 weeks.
  Interventions: Drug: Dose Level 1 ACU-D1 ointment; Procedure: Vulvar/ Perianal Biopsy
- Level 2 (Experimental): If there are no DLTs to Dose Level 1 then, 3 new study participants will proceed to Dose Level 2 at 5% ACU-D1.
  Interventions: Drug: Dose Level 2 ACU-D1 ointment; Procedure: Vulvar/ Perianal Biopsy
- Level 3 (Experimental): If there are no DLTs to Dose Level 2 then, 3 new study participants will proceed to Dose Level 3 at 10 % ACU-D1.
  Interventions: Drug: Dose Level 3 ACU-D1 ointment; Procedure: Vulvar/ Perianal Biopsy

INTERVENTIONS:
Drug: Dose Level 1 ACU-D1 ointment — ACU-D1 is a topical therapeutic agent that has pentaerythritol tetrakis (3-(3,5-di-tert-butyl-4-hydroxyphenyl) propionate) (PTTC) as its major active ingredient. PTTC is a novel proteasome inhibitor that has antiangiogenic and anti-inflammatory activities that reduce pro-inflammatory cytokines. ACU-D1 ointment contains a range of 2.5% to 10% weight by volume of PTTC.
  Level 1 will consist of 2.5% ACU-D1 ointment, used twice daily for 4 weeks.
  Arms: Level 1
Drug: Dose Level 2 ACU-D1 ointment — Level 2 will consist of 5% ACU-D1 ointment, used twice daily for 4 weeks.
  Arms: Level 2
Drug: Dose Level 3 ACU-D1 ointment — Level 3 will consist of 10% ACU-D1 ointment, used twice daily for 4 weeks.
  Arms: Level 3
Procedure: Vulvar/ Perianal Biopsy — 3 vulvar or perianal biopsies are to be performed at the screening as well as at the end of the study (week 4).

SUMMARY:
The goal of this study is to test the maximum tolerated dose of ACU-D1 in HIV-positive people with HPV-associated vulvar and perianal lesions. The main questions it aims to answer are:

* The maximum tolerated dose of ACU-D1
* Safety and tolerability of topical ACU-D1
* Whether topical ACU-D1 induces p53 and p53-mediated downstream signaling (including p21 induction) in HPV-related lesions
* Whether topical ACU-D1 enhances markers of immunity in HPV-infected HIV-positive individuals

Participants will be asked

* To apply ACU-D1 on the lesions twice daily for 4 weeks
* 3 biopsies will be performed at the screening and 3 at the end of 4 weeks.

DETAILED DESCRIPTION:
From 2016 to 2019, Georgia faced the highest incidence of HIV diagnosis among the fifty states ranging from 40.2 to 26.2 per 100,000 individuals. HIV-infected men and women living in the southern United States experience inadequate treatment services despite bearing the highest burden of new infections as the modern epicenter of the HIV epidemic. There has been considerable research on racial disparities and HIV incidence, but there is a paucity of data on differences in treatment outcomes, particularly those related to comorbidities.

HPV and HIV infection are the most significant risk factors for the development of High grade squamous intraepithelial lesion (HSIL), a documented precursor of cervical and anal cancer. While the mass availability of antiretroviral therapy has reduced the risk of AIDS-related deaths, it is estimated that over one-third of deaths within the HIV-infected population are a result of cancer. A number of these cancer deaths among people with HIV are attributable to the rising incidence of anogenital HPV infection within this population. Meta-analyses have documented a 28-fold and 6-fold higher risk of developing anal and cervical cancer, respectively, among PWH compared to the general population. African American individuals, men who have sex with men, and those residing in low-income areas, face a risk of non-AIDS-defining malignancies that extends beyond what can be explained by individual risk behaviors and coinfection. As the life expectancy of HIV-positive men and women approaches that of healthy individuals due to the success of antiretroviral treatment, there is a growing demand for a variety of anal and cervical cancer prevention methods amongst individuals with HIV.

HPV-associated cancer prevention efforts for people with HIV remain inadequate, particularly in low-resource settings. Health disparities by socioeconomic, ethnic, and gender identity groups are exacerbated by a lack of access to routine screening and treatment of vulvar and perianal premalignant disease. Moreover, few studies address the management and treatment of vulvar and perianal premalignant disease. This prompts extrapolation of treatment strategies from cervical premalignant disease, which are mainly ablative or excisional, and are thereby associated with higher risks for morbidity from treatment. Off-label topical treatment options, such as imiquimod and 5- 5-fluorouracil, have high side effect profiles (e.g., disfigurement and pain) when applied to the vulva and perianus, which prompt low compliance rates. Study participants may face multiple rounds of treatment with imiquimod or 5-fluorouracil due to high recurrence rates, further affecting compliance due to their negative side effect profiles. Also, imiquimod is cost-prohibitive for many members of our study population.

The development of a topical drug that has the potential to treat and reduce the volume of vulvar and perianal premalignant disease will widen the preventive treatment options in populations significantly burdened by vulvar and perianal cancers. ACU-D1 may address the unmet need for treatment of premalignant HPV-related anogenital disease among people living with HIV and others affected by this medical condition.

ACU-D1 is a topical therapeutic agent that has pentaerythritol tetrakis (3-(3,5-di-tert-butyl-4-hydroxyphenyl) propionate) (PTTC) as its major active ingredient. PTTC is a novel proteasome inhibitor that has antiangiogenic and anti-inflammatory activities that reduce pro-inflammatory cytokines. ACU-D1 ointment contains a range of 2.5% to 10% weight by volume of PTTC. The safety and efficacy of the ointment on facial skin have been validated in an FDA-approved trial for rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years and older
* HIV-infected
* Able to provide informed consent
* Biopsy-proven HSIL disease of the vulvar and perianal region with a total disease volume of 3 cm or greater
* Combined antiretrovirals (cART) adherence
* CD4 count > 200 cells/ml
* Sustained undetectable viral load for ≥ 3 months
* If applicable, on reliable birth control such as combined oral contraceptive pills (OCP), bilateral tubal ligation (BTL), a long-acting reversible contraceptive, or Depo-Provera (birth control shot)
* Willingness to conform to study requirements
* Reliable follow-up and contact information
* No risk factors or clinical suspicion for micro-invasive disease and absence of medical condition that interferes with the conduct of the study in the investigator's opinion

Exclusion Criteria:

* Currently pregnant (confirmed by collecting urine for HCG pregnancy test) or lactating

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of ACU-D1 | Baseline, week 4
  Subjects will be monitored during the trial for adverse events, tolerability and compliance using the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
  The dose level at which no more than 33% of study participants have a DLT will be considered the maximum tolerated dose.

SECONDARY OUTCOMES:
Ability of ACU-D1 to induce p53 and p21 in HPV lesions | Baseline, week 4
  The biopsies collected at the the 1st study visit and at the last study visit (week 4) mark will be examined using immunohistochemistry to determine gene activity and be used for other biomolecular assays
Safety of ACU-D1: Time of maximum observed concentration (tmax) | Before ointment application (0hr), 0.25 hour, 0.50 hour, 1hour, 1.5 hour, 2 hour, 4, 8 hour and 12 hour
  Pharmacokinetic studies will be performed on 3 participants after the 4th week of 10% ACU-D1 ointment application. As part of the studies, these 3 subjects will be admitted to the Grady satellite of the Atlanta Clinical and Translational Science Institute (ACTSI) where blood and urine samples will be collected in quick succession.
Safety of ACU-D1: Maximum concentration (Cmax) | Before ointment application (0hr), 0.25 hour, 0.50 hour, 1hour, 1.5 hour, 2 hour, 4, 8 hour and 12 hour
  Pharmacokinetic studies will be performed on 3 participants after the 4th week of 10% ACU-D1 ointment application. As part of the studies, these 3 subjects will be admitted to the Grady satellite of the Atlanta Clinical and Translational Science Institute (ACTSI) where blood and urine samples will be collected in quick succession.
Safety of ACU-D1: Area under the concentration-time curve for the last measurable concentration (AUC0-last) | Before ointment application (0hr), 0.25 hour, 0.50 hour, 1hour, 1.5 hour, 2 hour, 4, 8 hour and 12 hour
  Pharmacokinetic studies will be performed on 3 participants after the 4th week of 10% ACU-D1 ointment application. As part of the studies, these 3 subjects will be admitted to the Grady satellite of the Atlanta Clinical and Translational Science Institute (ACTSI) where blood and urine samples will be collected in quick succession.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Flowers, MD, MPH, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and analysis will be shared for publication purposes
Supporting Information: Study Protocol, SAP
Time Frame: After analyses have been completed